CLINICAL TRIAL: NCT00004876
Title: A Randomized Study Comparing Carboplatin and Thalidomide With Carboplatin Alone in Patients With Stage Ic - IV Ovarian Cancer
Brief Title: Carboplatin With or Without Thalidomide in Treating Patients With Ovarian Epithelial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Research UK (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000067536; ICRF-96.084; EU-99018
Record Dates: First submitted 2000-03-07; First posted 2003-01-27 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2011-11

CONDITIONS: Ovarian Cancer
Keywords: stage IV ovarian epithelial cancer; stage IC ovarian epithelial cancer; stage IIA ovarian epithelial cancer; stage IIB ovarian epithelial cancer; stage IIC ovarian epithelial cancer; stage IIIA ovarian epithelial cancer; stage IIIB ovarian epithelial cancer; stage IIIC ovarian epithelial cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Carboplatin; Thalidomide

INTERVENTIONS:
Drug: carboplatin
Drug: thalidomide

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Thalidomide may stop the growth of ovarian cancer by stopping blood flow to the tumor.

PURPOSE: This randomized phase II trial is studying how well giving carboplatin together with thalidomide works compared to carboplatin alone in treating patients with ovarian epithelial cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety of carboplatin and thalidomide in patients with stage IC-IV ovarian cancer.
* Determine the antiangiogenic effect of thalidomide in this patient population.
* Compare the efficacy of carboplatin with or without thalidomide in this patient population.

OUTLINE: This is a randomized study. Patients are randomized to one of two treatment arms.

* Arm I: Patients receive carboplatin IV over 1 hour. Treatment continues every 4 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive carboplatin as in arm I. Patients receive thalidomide orally once daily. Thalidomide treatment continues for up to 24 weeks commencing on the first day of carboplatin therapy and ceasing 4 weeks after the last course of carboplatin.

PROJECTED ACCRUAL: Approximately 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage IC-IV ovarian epithelial cancer
* Post-menopausal OR
* Prior bilateral salpingo-oophorectomy and/or total abdominal hysterectomy

PATIENT CHARACTERISTICS:

Age:

* Over 18

Performance status:

* WHO 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* No other concurrent invasive malignancies
* Not pregnant
* No diabetes mellitus
* No chronic neurological disease causing peripheral neuropathy

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No other concurrent cytotoxic agents

Endocrine therapy:

* Not specified

Radiotherapy:

* Concurrent local radiotherapy for treatment of secondary disease sites allowed

Surgery:

* See Disease Characteristics

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 1999-08

PRIMARY OUTCOMES:
Safety
Response
Markers of angiogenesis

CONTACTS AND LOCATIONS:
Overall Officials: T.S. Ganesan, MD, Study Chair — Oxford University Hospitals NHS Trust
Locations (1):
- Oxford Radcliffe Hospital, Oxford, England, United Kingdom

REFERENCES:
- [Result] Muthuramalingam SR, Braybrooke JP, Blann AD, Madhusudan S, Wilner S, Jenkins A, Han C, Kaur K, Perren T, Ganesan TS. A prospective randomised phase II trial of thalidomide with carboplatin compared with carboplatin alone as a first-line therapy in women with ovarian cancer, with evaluation of potential surrogate markers of angiogenesis. Eur J Gynaecol Oncol. 2011;32(3):253-8. PMID 21797111
- [Result] Muthuramalingam SR, Braybrooke JP, Madhusudan S, et al.: A randomised phase two study of carboplatin versus carboplatin and thalidomide in patients with ovarian cancer, with evaluation of potential surrogate markers of angiogenesis. [Abstract] Int J Gynecol Cancer 14 (Suppl 1): A-303, 86, 2004.